CLINICAL TRIAL: NCT02946047
Title: Pilot Study of Ixazomib to Reduce the Number of HIV DNA Positive Lymphoid Cells
Brief Title: The Effect of Ixazomib on the Latent HIV Reservoir
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Nathan W. Cummins, M.D., MD, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16-001938
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Results first posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Antiretroviral Therapy (ART)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ixazomib 1 mg (Experimental): Cohort A: Patients will receive ixazomib 1mg 3 times monthly for 12 weeks, then weekly for 12 weeks.
  Interventions: Drug: Ixazomib 1 MG
- Ixazomib 2 mg (Experimental): Cohort B: Patients will receive ixazomib 2mg 3 times monthly for 12 weeks, then weekly for 12 weeks.
  Interventions: Drug: Ixazomib 2 MG
- Ixazomib 3 mg (Experimental): Cohort C: Patients will receive ixazomib 3 mg 3 times monthly for 12 weeks, then weekly for 12 weeks.
  Interventions: Drug: Ixazomib 3 MG
- Ixazomib 4 mg (Experimental): Cohort D: Patients will receive ixazomib 4mg 3 times monthly for 12 weeks, then weekly for 12 weeks.
  Interventions: Drug: Ixazomib 4 MG

INTERVENTIONS:
Drug: Ixazomib 1 MG — 1 mg on days 1, 8 and 15 for three 28 days cycles, then be reviewed by DSMB and based upon their recommendation patients will receive ixazomib once weekly for 12 weeks or ixazomib 1 mg on days 1, 8 and 15 for three 28 days cycles. Visits 3-15 will have a window of ± 3 days.
  Other Names: Ninlaro
  Arms: Ixazomib 1 mg
Drug: Ixazomib 2 MG — 2mg on days 1, 8 and 15 for three 28 days cycles, then be reviewed by DSMB and based upon their recommendation patients will receive ixazomib once weekly for 12 weeks or ixazomib 2 mg on days 1, 8 and 15 for three 28 days cycles. Visits 3-15 will have a window of ± 3 days.
  Other Names: Ninlaro
  Arms: Ixazomib 2 mg
Drug: Ixazomib 3 MG — 3 mg on days 1, 8 and 15 for three 28 days cycles, then be reviewed by DSMB and based upon their recommendation patients will receive ixazomib once weekly for 12 weeks or ixazomib 3 mg on days 1, 8 and 15 for three 28 days cycles. Visits 3-15 will have a window of ± 3 days.
  Other Names: Ninlaro
  Arms: Ixazomib 3 mg
Drug: Ixazomib 4 MG — 4 mg on days 1, 8 and 15 for three 28 days cycles, then be reviewed by DSMB and based upon their recommendation patients will receive ixazomib once weekly for 12 weeks or ixazomib 4 mg on days 1, 8 and 15 for three 28 days cycles. Visits 3-15 will have a window of ± 3 days.
  Other Names: Ninlaro
  Arms: Ixazomib 4 mg

SUMMARY:
The primary purpose of the trial is to determine the safety and tolerability of ixazomib in HIV infected patients on antiretroviral therapy. The secondary purpose is to determine the effect of ixazomib on the size of the HIV reservoir.

ELIGIBILITY:
Inclusion Criteria:

* The following laboratory values obtained <=14 days prior to registration.
* ANC ≥ LLN (lower limit of normal) and ≤ULN (upper limit of normal), Hgb ≥ LLN and ≤ULN, PLT ≥ LLN and ≤ULN
* Total bilirubin ≤ULN and the direct bilirubin must be ≤ ULN; AST <1.5 x ULN and ALT <1.5 x ULN
* Creatinine <2.0 x ULN and an estimated creatinine clearance > 60 ml/min
* HIV infection with suppressed viral replication on at least 3 active drug ART for at least 6 months
* Suppressed viral replication is defined by plasma HIV viral load <20copies/mL.
* Patient must have HIV viral load <20 copies/ml on two occasions at least 3 months apart.
* In the opinion of the treating physician, patients must have available other regimens likely to suppress HIV should their current regimen fail.
* Male or female patients age >=18 years
* A plasma HIV RNA viral load demonstrating a measure of <20 copies/mL within 30 days prior to study initiation.
* CD4 count >500 cells/mm3 within 30 days prior to study enrollment
* Females must have a negative pregnancy test prior to receiving the 1st dose of ixazomib and be postmenopausal for at least 1 year before the screen visit, or surgically sterile,
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception AND a second method of contraception for female partners of childbearing potential during the entire study treatment period and through 90 days after the last dose of ixazomib,
  * OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
  * AND
  * Agree to forego sperm donation for the same period as above.

Exclusion Criteria:

* The following laboratory values obtained <=14 days prior to registration.

  * ANC < LLN and >ULN, Hgb < LLN and >ULN, PLT < LLN and >ULN
  * Total bilirubin >ULN or the direct bilirubin is > ULN; AST >1.5 x ULN or AST >1.5 x ULN
  * Creatinine >=2.0 x ULN or an estimated creatinine clearance <=60mL/min
* Diagnosed and treated for a malignancy within 5 years before randomization, or previously diagnosed with a malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Any infection except HIV (excluding benign conditions that is unlikely to be affected or modulated by treatment with ixazomib, e.g. stye or furuncle), or treatment with anti-infective agents within 14 days of enrollment.
* Pregnant women
* Women of childbearing potential and Nursing women
* Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse, while taking the drug and for 90 days after stopping ixazomib.
* Any history of peripheral neuropathy, or peripheral neuropathy detected during the screening period.
* Major surgery within 14 days before study registration
* Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin,carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
* Evidence of current uncontrolled cardiovascular conditions, including serious cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months.
* QTc > 450 milliseconds (msec) for men and >470 milliseconds for women (83) on a 12 lead ECG obtained during the Screening period.
* Known hepatitis B DNA positive status and/or HBsAg positive and/or HBeAg positive, or active hepatitis C replication (HCV RNA positive) or currently on hepatitis C treatment.
* Known history of cirrhosis or active liver inflammation, including "fatty liver" or non-alcohol steatohepatitis (NASH).
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues or excipients in the various formulations.
* Any other recent or concurrent medical condition that, in the Investigator's opinion, would impose any risk to the patient
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Cummins, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixazomib 1 mg | Ixazomib 2 mg | Ixazomib 3 mg | Ixazomib 4 mg
Started | 4 | 3 | 3 | 7
Completed | 3 | 3 | 3 | 7
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixazomib 1 mg | Ixazomib 2 mg | Ixazomib 3 mg | Ixazomib 4 mg | Total
Number analyzed (Participants) | 4 | 3 | 3 | 7 | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.1 [49.9 to 58.2] | 49.3 [40.9 to 52.3] | 51.0 [39.3 to 53.5] | 49.0 [41.2 to 52.0] | 51.0 [45.1 to 55.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1
  Male | 4 | 3 | 3 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Number of treatment-emergent adverse events experienced by subjects as defined by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib 1 mg | Ixazomib 2 mg | Ixazomib 3 mg | Ixazomib 4 mg
Number analyzed (Participants) | 4 | 3 | 3 | 7
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Cell Associated HIV DNA in CD4 T Cell Subsets
Description: HIV copies per million CD4 T cells
Time Frame: 24 weeks
Population: 24 week data for 1 participant in the Ixazomib 1 mg arms was not collected or analyzed
Measure: Median (Inter-Quartile Range); unit: copies per million
Arm/Group | Ixazomib 1 mg | Ixazomib 2 mg | Ixazomib 3 mg | Ixazomib 4 mg
Number analyzed (Participants) | 4 | 3 | 3 | 7
copies per million
  Baseline | 378 [208 to 837] | 626 [54 to 1385] | 664.8 [130 to 1014] | 416 [39 to 988]
  24 weeks: number analyzed (Participants) | 3 | 3 | 3 | 7
  24 weeks | 394 [137 to 812] | 425 [45 to 1715] | 624 [98 to 1125] | 481 [24 to 846]

3. Secondary Outcome: Culturable HIV by Quantitative Viral Outgrowth Assay
Description: Infectious units per million CD4 T cells
Time Frame: 24 weeks
Population: 24 week data for 1 participant in the Ixazomib 1 mg arms was not collected or analyzed
Measure: Median (Inter-Quartile Range); unit: units per million
Arm/Group | Ixazomib 1 mg | Ixazomib 2 mg | Ixazomib 3 mg | Ixazomib 4 mg
Number analyzed (Participants) | 4 | 3 | 3 | 7
units per million
  Baseline | 0.49 [0.15 to 1.23] | 0.30 [0.14 to 1.60] | 0.62 [0.30 to 2.12] | 1.54 [0.15 to 2.95]
  24 weeks: number analyzed (Participants) | 3 | 3 | 3 | 7
  24 weeks | 0.30 [0.30 to 0.66] | 0.48 [0.10 to 0.65] | 0.82 [0.81 to 1.07] | 1.31 [0.10 to 2.58]

4. Secondary Outcome: Absolute CD4 T Cell Count
Description: Cells per microliter
Time Frame: 24 weeks
Population: 24 week data for 1 participant in the Ixazomib 1 mg arms was not collected or analyzed
Measure: Median (Inter-Quartile Range); unit: cells/mmˆ(3)
Arm/Group | Ixazomib 1 mg | Ixazomib 2 mg | Ixazomib 3 mg | Ixazomib 4 mg
Number analyzed (Participants) | 4 | 3 | 3 | 7
cells/mmˆ(3)
  Baseline | 724 [676 to 830] | 914 [790 to 968] | 1130 [1029 to 1240] | 735 [680 to 770]
  24 weeks: number analyzed (Participants) | 3 | 3 | 3 | 7
  24 weeks | 714 [696 to 735] | 809 [771 to 813] | 765 [676 to 825] | 632 [548 to 768]

5. Secondary Outcome: Absolute CD8 T Cell Count
Description: Cells per microliter
Time Frame: 24 weeks
Population: 24 week data for 1 participant in the Ixazomib 1 mg arms was not collected or analyzed
Measure: Median (Inter-Quartile Range); unit: cells/mmˆ(3)
Arm/Group | Ixazomib 1 mg | Ixazomib 2 mg | Ixazomib 3 mg | Ixazomib 4 mg
Number analyzed (Participants) | 4 | 3 | 3 | 7
cells/mmˆ(3)
  Baseline | 508 [504 to 810] | 803 [716 to 834] | 1014 [868 to 1208] | 573 [405 to 712]
  24 weeks: number analyzed (Participants) | 3 | 3 | 3 | 7
  24 weeks | 387 [337 to 428] | 885 [624 to 888] | 689 [573 to 723] | 416 [332 to 486]

6. Secondary Outcome: CD4/CD8 Ratio
Description: CD4/CD8 T cell count ratio
Time Frame: 24 weeks
Population: 24 week data for 1 participant in the Ixazomib 1 mg arms was not collected or analyzed
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Ixazomib 1 mg | Ixazomib 2 mg | Ixazomib 3 mg | Ixazomib 4 mg
Number analyzed (Participants) | 4 | 3 | 3 | 7
ratio
  Baseline | 1.45 [1.10 to 1.67] | 1.14 [0.95 to 1.38] | 1.28 [1.04 to 1.31] | 1.58 [1.15 to 1.82]
  24 weeks: number analyzed (Participants) | 3 | 3 | 3 | 7
  24 weeks | 1.84 [1.64 to 2.24] | 0.92 [0.87 to 1.57] | 1.17 [1.01 to 1.42] | 1.75 [1.42 to 2.09]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 7 months on all participatns.
Arm/Group | Ixazomib 1 mg | Ixazomib 2 mg | Ixazomib 3 mg | Ixazomib 4 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/7
Other Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 1/3 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib 1 mg (N=4) | Ixazomib 2 mg (N=3) | Ixazomib 3 mg (N=3) | Ixazomib 4 mg (N=7)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Edema Limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT02946047/Prot_SAP_000.pdf